CLINICAL TRIAL: NCT06760520
Title: A Single-arm, Prospective, Phase II Clinical Study of Short-course Radiotherapy Followed by CAPOX and Ivonescimab for Locally Advanced Low-middle Rectal Cancer with a High Risk of Recurrence
Brief Title: Short-course Radiotherapy Followed by CAPOX and Ivonescimab for Locally Advanced Rectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Yugui Lian, Clinical Professor, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-KY-1578-002
Record Dates: First submitted 2024-12-21; First posted 2025-01-07 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Locally Advanced Rectal Cancer
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ivonescimab+chemotherapy (Experimental): Local advanced rectal cancer with short-course radiotherapy followed by sequential chemotherapy and ivonescimab
  Interventions: Drug: Ivonescimab (SMT112 or AK112) Injection

INTERVENTIONS:
Drug: Ivonescimab (SMT112 or AK112) Injection — Eligible subjects will receive short-course radiotherapy (SCRT), 25Gy/5f/1 week. 1-2 weeks after the end of treatment, subjects continued to receive neoadjuvant chemotherapy combined with immunotherapy regimen for 4 cycles: AK112 20 mg/kg, intravenous infusion every 3 weeks (Q3W), plus CAPOX (capecitabine: 850-1000mg/m2, bid, po, d1-14, oxaliplatin: 130mg/m2, ivgtt, d1), Q3W. Neoadjuvant therapy was assessed 2 weeks after the end of neoadjuvant therapy, and TME surgery was performed 4 weeks after the end of neoadjuvant therapy (R0 surgery was performed).

SUMMARY:
This study is a single-arm, prospective, phase II clinical study to evaluate the efficacy and safety of preoperative short-course radiotherapy combined with ivonescimab and chemotherapy + total mesorectal excision(TME) surgery in patients with advanced rectal cancer.

DETAILED DESCRIPTION:
Studies included a screening period (no more than 28 days after participants signed informed consent form to 28 days before first dose), treatment (receiving appropriate treatment until disease progression, intolerable toxicity, withdrawal of informed consent, death or study end, whichever occurs first), and follow-up (including safety follow-up and survival follow-up).

Eligible subjects will receive short-course radiotherapy (SCRT), pelvic 25Gy/5f/1 week. 1-2 weeks after the end of treatment, subjects continued to receive neoadjuvant chemotherapy combined with immunotherapy regimen for 4 cycles: ivonescimab 20 mg/kg, intravenous infusion every 3 weeks (Q3W), plus CAPOX (capecitabine: 850-1000mg/m2, bid, po, d1-14, oxaliplatin: 130mg/m2, ivgtt, d1), Q3W. Neoadjuvant therapy was assessed 2 weeks after the end of neoadjuvant therapy, and TME surgery was performed 4 weeks after the end of neoadjuvant therapy (R0 surgery was performed). Patients can choose to enter the organ preservation observation; If the efficacy after preoperative chemoradiotherapy is evaluated as clinical complete remission (cCR) and the patient strongly refuses surgery, the patient should be informed of the risk of recurrence and ask the patient to sign a rejection of surgery. Medication safety is assessed and, depending on the severity of adverse events (AEs) and drug relevance, investigators will take steps to ensure subject safety. After surgery (or patients who strongly refuse surgery) there is a 30- and 90-day safety follow-up, and survival assessments are performed every 3 months to obtain survival information and collect new tumor treatment information until the death of the participant, withdrawal of informed consent, or the end of the study, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* ECOG score of 0-1;
* histologically or cytologically confirmed colorectal adenocarcinoma with non-distant metastasis
* Tumor distance from anal verge ≦10cm
* at least one high-risk criterion defined by pelvic MRI: cT stage >T2 (tumor invades intrinsic muscularis propria by more than 5 mm); Extramural vascular invasion; cN2; Involvement of the rectal mesorectal fascia (tumor or lymph node ≤1mm from the rectal mesorectal fascia); Lateral lymph node short diameter ≥5mm
* enough organ function

Exclusion Criteria:

* with known MSI-H or dMMR
* Multiple primary adenocarcinomas
* History of pelvic radiotherapy
* Previous immunotherapy, including immune checkpoint inhibitors (e.g., anti-PD-1 antibody, anti-PD-L1 antibody, anti-CTLA-4 antibody, etc.), immune checkpoint agonists (e.g., ICOS, CD40, CD137, GITR, OX40 antibody, etc.), immunocellular therapy, and other treatments targeting the immune mechanism of the tumor.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2027-12-20 (Estimated); Study Completion 2031-12-20 (Estimated)

PRIMARY OUTCOMES:
Complete response rate (CR, pCR plus cCR ) | pCR rate : within 1 week after surgery；cCR：12-13 weeks after radiotherapy ends
  pathological complete response rate plus clinical complete response rate

SECONDARY OUTCOMES:
3-years DFS rate | From date of treatment until the date of first documented disease relapse or date of death from any cause, whichever came first about 3years.
5-years OS rate | From date of treatment until date of death from any cause,about 5 years
ORR | up to 2 years
  objective response rate
Incidence and severity of adverse events (AEs) | up to 2 years
Tumor downstaging rate | up to 2 years
2-year organ preservation observation rate | up to two years
surgical complication | 30 days after surgery